CLINICAL TRIAL: NCT01835782
Title: Determining the Safety of L-Serine in Subjects With Amyotrophic Lateral Sclerois (ALS) at Varied Doses.
Brief Title: Determining the Safety of L-serine in ALS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Phoenix Neurological Associates, LTD (Other)
Collaborators: Institute for Ethnomedicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L-Serine2013; IND (Other: 116871)
Record Dates: First submitted 2013-03-27; First posted 2013-04-19 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ALS; L-Serine; BMAA
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Serine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2.5 grams BID (Active Comparator): 5 Patients will be evenly randomized into this group
  Interventions: Drug: L-Serine
- .5 grams BID (Active Comparator): 5 Patients will be evenly randomized into this group
  Interventions: Drug: L-Serine
- 7.5 grams BID (Active Comparator): 5 Patients will be evenly randomized into this group
  Interventions: Drug: L-Serine
- 15 grams BID (Active Comparator): 5 Patients will be evenly randomized into this group
  Interventions: Drug: L-Serine

INTERVENTIONS:
Drug: L-Serine

SUMMARY:
The purpose of this study is to determine the safety of L-Serine in subjects with Amyotrophic Lateral Sclerosis (ALS) at varied doses.

DETAILED DESCRIPTION:
Previous studies into the Guamian ALS-Parkinson's Dementia complex has identified β-methylamino-L-alanine (BMAA), as a potential neurotoxin responsible for this disease. BMAA is a non-essential amino acid and is produced by a cyanobacterium which is present in all ecosystems. Subsequently several groups have identified high concentrations of BMAA in brain tissues of patients from North America and Europe with several neurodegenerative diseases including ALS, Parkinson's Disease and Alzheimer's Diseases. It has been hypothesized that chronic intake of BMAA in the diet leads to mis-incorporation of the amino acid into brain proteins, where it produces slow neuronal damage and recent evidence has shown that BMAA is mis-incorporated into proteins in neuronal cell lines via seryl tRNA synthetase, thereby producing protein mis-folding and protein aggregates, leading to cell death. It has been demonstrated in mammalian neuronal cell cultures that exogenous L-serine could prevent the BMAA neurotoxin from being mis-incorporated into proteins, thereby preventing cell death and that very high doses of L-serine may compete with the transport of a number of non-essential amino acids across the blood-brain barrier via the y+ transporter. These findings have led us to believe that high doses of L-serine could possibly stop the mis-incorporation of BMAA into brain proteins which in turn would slow or even abate the progression of ALS. This study will determine the safety of different doses of L-serine given to ALS subjects at 0.5 gm twice daily (BID), 2.5gm BID, 7.5g BID or 15 grams BID for six months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Male or Female
3. Clinically diagnosed with probable or definite ALS based on El Escorial criteria
4. ALSFRS-R > 25
5. Able to provide informed consent to and comply with all medical procedures

Exclusion Criteria:

1. Outside age range of 18-85
2. Subjects with forced vital capacity (FVC) below 60%
3. Evidence of any motor neuron disease for over 3 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Safety of L-Serine | 1-6 months
  Determining the safety of L-Serine given at 0.5 gm twice daily (BID), 2.5gm BID, 7.5g BID or 15 grams BID for six months by assessing the total number of adverse events (AE)during treatment

SECONDARY OUTCOMES:
Measure levels of β-Methylamino-L-alanine (BMAA) in blood, urine and Cerebrospinal fluid (CSF) to determine if there is a decline in levels over the course of treatment | 1-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Levine, MD, Principal Investigator — Phoenix Neurological Associates, LTD
Locations (2):
- United States (2):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - Forbes Norris MDA/ALS Research Center, San Francisco, California